CLINICAL TRIAL: NCT00986089
Title: Pilot Study of Copper IUD Placement at the Time of Cesarean Section
Brief Title: Intrauterine Device (IUD) Placement at the Time of Cesarean Section
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left the University of Kentucky before enrollment could begin.
Sponsor: University of Kentucky (Other)
Collaborators: Duramed Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 08-0938-F6A
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2013-08

CONDITIONS: Intrauterine Device Placement
Keywords: post-placental; IUD; Copper IUD; cesarean section; immediate post-partum; continuation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women who have an IUD placed at the time of c-section

SUMMARY:
To evaluate the continuation of the Copper IUD at one year after placement through the cesarean incision into the uterus at the time of cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Desire an IUD post-partum and are willing to use the copper IUD.
* They will also need to be patients at one of our OBGYN clinics at the university of Kentucky.

Exclusion Criteria:

* Post-partum hemorrhage,
* Chorioamnionitis (or a fever >101 at the time of cesarean),
* Women on antibiotic or immunosuppressive therapies,
* Cervical dilation > 5 cm at the time of c-section, OR
* Excessive intraoperative blood loss.
* Also women with contraindications to a copper IUD: Wilson's disease, unusual uterine shape or known uterine anomaly.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women ages 18-40 who are undergoing a scheduled cesarean section, or women who are attempting to VBAC and want an IUD post partum will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Continuation at one year | 1 year

SECONDARY OUTCOMES:
satisfaction with placement at time of cesarean | 4-6 months and 1 year
bleeding profile | 6 months

REFERENCES:
- [Background] Hayes JL, Cwiak C, Goedken P, Zieman M. A pilot clinical trial of ultrasound-guided postplacental insertion of a levonorgestrel intrauterine device. Contraception. 2007 Oct;76(4):292-6. doi: 10.1016/j.contraception.2007.06.003. Epub 2007 Aug 6. PMID 17900440
- [Background] Liu BH, Zhang LY, Zhang BR. Intrauterine contraceptive device insertion with suture fixation at cesarean section. Chin Med J (Engl). 1983 Feb;96(2):141-4. PMID 6406171
- [Background] Eroglu K, Akkuzu G, Vural G, Dilbaz B, Akin A, Taskin L, Haberal A. Comparison of efficacy and complications of IUD insertion in immediate postplacental/early postpartum period with interval period: 1 year follow-up. Contraception. 2006 Nov;74(5):376-81. doi: 10.1016/j.contraception.2006.07.003. Epub 2006 Sep 15. PMID 17046378